CLINICAL TRIAL: NCT05781698
Title: Repurposing Fenofibrate in Modulating mTOR/NLRP3 Inflammasome in Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Manal Ali Mahrous Hamouda Faculty of Pharmacy, Menufia University (Unknown)
Responsible Party: Principal Investigator, Mostafa Bahaa, Teaching Assistant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-2023
Record Dates: First submitted 2023-03-11; First posted 2023-03-23 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Mesalamine; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The control group ( Mesalamine group, n =35 ) will receive 1 g mesalamine three times daily for 6 months
  Interventions: Drug: Mesalamine
- Fenofibrate group (Active Comparator): Patients will receive 1 g mesalamine three times daily plus Fenofibrate (160 mg/day) for 6 months
  Interventions: Drug: Mesalamine; Drug: Fenofibrate

INTERVENTIONS:
Drug: Mesalamine — mesalamine is the cornerstone used for the treatment of mild to moderate ulcerative colitis
Drug: Fenofibrate — Fibrates, which are specific pharmacological agonists of PPARα, have been widely used in the treatment for hypercholesterolemia and hypertriglyceridemia
  Arms: Fenofibrate group

SUMMARY:
Fibrates, specific pharmacological agonists of PPARα, have been widely used to treat hypercholesterolemia and hypertriglyceridemia. Apart from their metabolic action, anti-inflammatory properties of fibrates have been described, including inhibition of NF-kappa B signaling and pro-inflammatory cytokine production. 4 Fenofibrate, an important peroxisome proliferator-activated receptor-a (PPAR- α) agonist, is widely used in clinical as a triglyceride (TG)-lowering agent

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years Both male and female will be included Negative pregnancy test and effective contraception. Mild and moderate UC patients diagnosed and confirmed by endoscope

Exclusion Criteria:

Breast feeding Significant liver and kidney function abnormalities Colorectal cancer patients Other inflammatory bowel diseases (CD). Patients with severe UC Patients taking rectal or systemic steroids Patients taking immunosuppressives or biological therapies Addiction to alcohol and/or drugs Known allergy to the Fenofibrate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
• The primary endpoint is the change in disease activity index and the improvement in health-related quality of life (HRQL). | 6 months
  • The primary endpoint is the change in disease activity index and the improvement in health-related quality of life (HRQL).

SECONDARY OUTCOMES:
The secondary endpoint is estimated by changes in serum biomarkers. | 6 months
  The secondary endpoint is estimated by changes in serum biomarkers such as adenosine monophosphate activated protein kinase

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Menoufia University, Tanta, Shebeen El-Kom, Egypt

REFERENCES:
- [Derived] Alarfaj SJ, Bahaa MM, Elmasry TA, Elberri EI, El-Khateeb E, Hamouda AO, Salahuddin MM, Kamal M, Gadallah AA, Eltantawy N, Yasser M, Negm WA, Hamouda MA, Alsegiani AS, Alrubia S, Eldesoqui M, Abdallah MS. Fenofibrate as an Adjunct Therapy for Ulcerative Colitis: Targeting Inflammation via SIRT1, NLRP3, and AMPK Pathways: A Randomized Controlled Pilot Study. Drug Des Devel Ther. 2024 Nov 16;18:5239-5253. doi: 10.2147/DDDT.S490772. eCollection 2024. PMID 39575188